CLINICAL TRIAL: NCT05627817
Title: Timing of Preload Responsiveness in Sepsis and Septic Shock
Brief Title: Timing of Preload Responsiveness in Sepsis
Acronym: TIPRES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Principal Investigator, Bicetre Hospital
Other Study IDs: 2018-A03040-55
Record Dates: First submitted 2022-11-15; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Septic Shock; Fluid Responsiveness
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During acute circulatory failure, volume expansion does not always lead to a significant increase in cardiac output (fluid responsiveness). After initial resuscitation by rapid fluid administration, cardiac preload is no longer extremely low and only half of the patients respond to further volume expansion with the expected increase in cardiac output (fluid unresponsiveness). However, the time delay or the volume of fluid needed to be administered from the state of fluid responsiveness to fluid unresponsiveness is still not determined.

Objective To determine, in critically ill patients with acute circulatory failure,

1. : the time and/or the volume of fluid needed from the state of fluid responsiveness to fluid unresponsiveness during septic shock.
2. : determine the factors that influence this time and volume.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Onset of septic shock

Exclusion Criteria:

* Planned to transfer the patient to another healthcare facility (inability to continue cardiac output measurements); urgent operation; Inability to measure the cardiac output.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who just arrive at the Intensive Care Unit (ICU) for septic shock need to be quickly resuscitated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The time delay from the state of fluid responsiveness to fluid unresponsiveness | 60 minutes after the evaluation of fluid responsiveness
  At the time of inclusion, the investigators use the tests available (fluid challenge, passive leg raising, end-expiratory occlusion test) to evaluate the presence of fluid responsiveness, and after one hour, the investigators repeat the test and to re-evaluate the presence of fluid responsiveness until the patient is no longer present the fluid responsiveness.
The volume of fluid needed from the state of fluid responsiveness to fluid unresponsiveness | 15-30 minutes during the fluid administration
  If the fluid challenge is performed, the volume of each time for the fluid administration should be noted until the patient is no longer fluid-responsive, then the investigators can calculate the total amount of the fluid administrated.

SECONDARY OUTCOMES:
The risk factors for the time delay | Through study completion, an average of 1 year
  Determine the factors that may influence the time delay from the state of fluid responsiveness to fluid unresponsiveness
The risk factors for the volume of fluid needed from the state of fluid responsiveness to fluid | Through study completion, an average of 1 year
  Determine the factors that may influence the volume of fluid administrated from the state of fluid responsiveness to fluid unresponsiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Bicetre Hospital, Paris, Val-de-Marne, France

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Monnet X, Teboul JL. My patient has received fluid. How to assess its efficacy and side effects? Ann Intensive Care. 2018 Apr 24;8(1):54. doi: 10.1186/s13613-018-0400-z. PMID 29691755
- [Background] Monnet X, Shi R, Teboul JL. Prediction of fluid responsiveness. What's new? Ann Intensive Care. 2022 May 28;12(1):46. doi: 10.1186/s13613-022-01022-8. PMID 35633423
- [Background] Roger C, Zieleskiewicz L, Demattei C, Lakhal K, Piton G, Louart B, Constantin JM, Chabanne R, Faure JS, Mahjoub Y, Desmeulles I, Quintard H, Lefrant JY, Muller L; AzuRea Group. Time course of fluid responsiveness in sepsis: the fluid challenge revisiting (FCREV) study. Crit Care. 2019 May 16;23(1):179. doi: 10.1186/s13054-019-2448-z. PMID 31097012
- [Background] Kattan E, Ospina-Tascon GA, Teboul JL, Castro R, Cecconi M, Ferri G, Bakker J, Hernandez G; ANDROMEDA-SHOCK Investigators. Systematic assessment of fluid responsiveness during early septic shock resuscitation: secondary analysis of the ANDROMEDA-SHOCK trial. Crit Care. 2020 Jan 23;24(1):23. doi: 10.1186/s13054-020-2732-y. PMID 31973735